CLINICAL TRIAL: NCT06293690
Title: Efficacy and Safety of Toripalimab Combined With SBRT in the Neoadjuvant Treatment for Operable or Potentially Operable Non-small Cell Lung Cancer in Stage IIA to IIIB
Brief Title: Toripalimab Combined With SBRT for NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Deping Zhao, Administrative Director of Thoracic Surgery, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L23-407
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non-small Lung Cancer
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT combined with immunochemotherapy (Other): A: Patients received preoperative neoadjuvant therapy: SBRT 12Gy on the first day, and Toripalimab (IV 240mg, q3W) combined with platinum-containing dual drugs on the second day. Two cycles in total.
  Interventions: Drug: Toripalimab
- SBRT combined with immunotherapy (Other): B:Patients received preoperative neoadjuvant therapy: SBRT 12Gy on the first day, and Toripalimab (IV 240mg, q3) on the second day. Two cycles in total.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Patients received preoperative neoadjuvant therapy: SBRT 12gy on the first day, and Toripalimab (iv 240mg, q3W) combined with platinum-containing dual drugs on the second day. Two cycles in total.
  Other Names: SBRT; platinum-containing dual drugs
  Arms: SBRT combined with immunochemotherapy
Drug: Toripalimab — Patients received preoperative neoadjuvant therapy: SBRT 12gy on the first day, and Toripalimab (iv 240mg, q3W) on the second day. Two cycles in total.
  Other Names: SBRT
  Arms: SBRT combined with immunotherapy

SUMMARY:
This study aimed to evaluate the efficacy and safety of Toripalimab injection (js001) combined with SBRT radiotherapy and neoadjuvant therapy with or without chemotherapy for operable or potentially operable stage IIa to IIIb NSCLC

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 75 years old, regardless of gender;
2. ECOG behavior status score 0-1 points;
3. Non small cell lung cancer diagnosed pathologically and clinically classified as stage IIA-IIIB (8th AJCC staging standard);
4. Sufficient tumor tissue can be provided for biomarker analysis;
5. Patients with distant metastasis are excluded through CT or PET/CT, and their physical condition is evaluated as acceptable for radical lung cancer surgery;
6. Primary lung lesions are suitable for SBRT treatment;
7. Confirming the absence of EGFR/ALK/ROS-1 sensitive gene mutations through molecular pathological diagnosis of the organization;
8. The main organ functions within 7 days before the first administration meet the following standards:

a Bone marrow function: hemoglobin ≥ 10.0 g/dL (no blood transfusion received within 28 days before hemoglobin test), absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L (no platelet transfusion or IL-11 treatment received within 14 days prior to platelet count test);b Coagulation function: INR and PT<1.5 × ULN, APTT ≤ 1.5 × ULN;c Liver function: transaminases (ALT and AST) ≤ 2.5 × ULN; Total bilirubin ≤ 1.5 × ULN (total bilirubin ≤ 2.5 in subjects with Gilbert's syndrome or liver metastasis) × ULN);d Renal function: serum creatinine clearance rate ≥ 60 mL/min (calculated according to Cockcroft Fault formula);e Adequate lung function: According to the doctor's judgment, lung function can meet the requirements of thymectomy surgery.

Exclusion Criteria:

1. Pathological findings indicate complex small cell lung cancer, etc;
2. History of previous lobectomy surgery and previous experience with radiotherapy and chemotherapy;
3. Patients with concurrent secondary primary cancer and a history of malignant tumors less than 5 years (excluding completely cured cervical carcinoma in situ or basal or squamous cell skin cancer);
4. The patient has any active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism, etc.);
5. Have active infection or active tuberculosis history requiring systemic treatment;
6. Those who have combined the following active infectious diseases, including those who are highly positive for hepatitis, known human immunodeficiency virus (HIV) infections, and sexually transmitted diseases such as active syphilis;
7. Those who are known to have or combine with other uncontrollable diseases and are unable to receive surgical treatment;
8. Physical examination or clinical trial findings that researchers believe may interfere with the results or increase the risk of treatment complications for patients;
9. Previous history of interstitial lung disease, drug-induced interstitial disease, or any clinically proven active interstitial lung disease, baseline CT scan reveals the presence of idiopathic pulmonary fibrosis; Uncontrolled large amounts of pleural or pericardial effusion;
10. Unstable systemic comorbidities (active infection period, moderate to severe chronic obstructive pulmonary disease, poorly controlled hypertension, unstable angina, congestive heart failure, myocardial infarction occurring within 6 months, severe mental disorders requiring drug control, metabolic diseases of the liver, kidney or other organs, neuropsychiatric disorders such as Alzheimer's disease);
11. History of congenital or acquired immunodeficiency diseases or organ transplantation;
12. Have received any of the following treatments:a Previously received chemotherapy, anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs, or other drugs that synergistically inhibit T cell receptors such as CTLA-4, OX-40, and CD137; Received any investigational medication within 4 weeks prior to the first use of the investigational medication;b Simultaneously enroll in another clinical study, unless it is an observational (non-intervention) clinical study or an intervention clinical study follow-up;c Individuals who have received anti-tumor vaccines or have received live vaccines within 4 weeks prior to the first administration of the investigational drug;d Having undergone major surgery or severe trauma within 4 weeks before the first use of the investigational drug;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Major pathological remission rate | 30 day
  The percentage of residual live tumor cells in the tumor bed after neoadjuvant therapy is ≤ 10%, regardless of whether there are residual live tumor cells in the lymph nodes.

SECONDARY OUTCOMES:
Complete pathological remission rate | 30 day
  After a complete evaluation of excised lung cancer specimens, including lymph nodes in all sampling areas, there was a lack of any surviving tumor cells when re examining HE slides
disease-free survival（DFS） | 3 years
  The time interval between receiving surgical treatment and tumor recurrence or death due to tumor progression
overall survival | 3 years
  The time interval between receiving surgical treatment and the patient's death due to any reason, and the patient is still alive during the final follow-up, with the survival time ending at the last follow-up.

OTHER OUTCOMES:
Adverse events | 24 hours
  Adverse events (AEs) related to the investigational drug, laboratory test outliers, and serious adverse events (SAEs) determined according to the NCI-CTCAE V5.0 standard

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No